CLINICAL TRIAL: NCT01085266
Title: HORIZON-Plus: An Open-Label Extension of the HORIZON Protocol (DIM20) Evaluating the Safety of Dimebon (Latrepirdine) in Subjects With Huntington Disease
Brief Title: An Extension of the HORIZON Protocol Evaluating the Safety of Dimebon (Latrepirdine) in Subjects With Huntington Disease
Acronym: HORIZON PLUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM20EXT
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — latrepirdine

ARMS (1):
- Dimebon (latrepirdine) (Experimental): Patients receive dimebon 10mg orally 3 times per day for 1 week and 20 mg orally 3 times per day thereafter.
  Interventions: Drug: Dimebon (latrepirdine)

INTERVENTIONS:
Drug: Dimebon (latrepirdine)

SUMMARY:
An open-label extension study of the HORIZON protocol evaluating the safety of dimebon (latrepirdine)in subjects with Huntington disease.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of 26 weeks of blinded treatment in the HORIZON study

Exclusion Criteria:

* Any other medical illness or unstable medical condition that may interfere with their ability to comply with study procedures and abide by study restrictions, or may interfere with the ability to interpret safety information.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual)